CLINICAL TRIAL: NCT01304862
Title: Electronic Self-management Resource Training for Mental Health
Acronym: eSMART-MH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Melissa D. Pinto-Foltz, KL2 SCHOLAR, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KL2RR024990 (NIH)
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Depression; Generalized Anxiety Disorder
MeSH Terms: conditions — Depression; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Self-management intervention (Experimental)
  Interventions: Behavioral: eSMART-MH intervention
- Educational Videos about Healthy Living (Active Comparator)
  Interventions: Behavioral: Educational videos about healthy living

INTERVENTIONS:
Behavioral: eSMART-MH intervention — Involves simulated interactions between participants and the virtual health care providers (avatars).
  Arms: Self-management intervention
Behavioral: Educational videos about healthy living — 20 minute screen-based educational videos on topics about healthy living--nutrition, physical activity, and sleep hygiene.
  Arms: Educational Videos about Healthy Living

SUMMARY:
The purpose of this study is to determine whether mental health treatment disengagement may be mitigated by reducing barriers to self-management and enhancing self-management skills.

DETAILED DESCRIPTION:
Each year, more than four million young adults (age 18-25 years old) in the U.S. receive psychotropic medication or psychotherapy as treatment for a mental illness. One in every four of these young adults will disengage from mental health treatment before significant symptom remission is achieved. Mental health treatment disengagement may be mitigated by reducing barriers to self-management and enhancing self-management skills. Electronic self-management resource training for mental health (eSMART-MH) is an innovative use of avatars-virtual persons who tailor responses to users-to improve mental health treatment disengagement.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of a diagnosis depression or generalized anxiety disorder greater than six months
* Young adults 18-25 years of age
* Prescribed psychotropic medication and/or psychotherapy
* Have a documented domestic telephone number
* Able to read and understand English

Exclusion Criteria:

* Participation in the eSMART-HD parent project

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-02; Primary Completion 2013-07-01 (Actual); Study Completion 2013-07-01 (Actual)

PRIMARY OUTCOMES:
Engagement in Mental Health Treatment: Medical Adherence Medication Module (MAMMM) | 12 weeks
  Medical Adherence Measure Medication Module (MAMMM) is a 7-item scale that will determine the patient's degree of engagement and initiation of mental health treatment.

SECONDARY OUTCOMES:
Mental Illness Stigma: Alienation Subscale | 12 weeks
  A 6-item four point Likert type scale that asks participants to rate each item from 1 (strongly disagree) to 4 (strongly agree); a higher score indicates more mental illness stigma.
Mental Health Literacy: In Our Own Voice Knowledge Measure (IOOVKM) | 12 weeks
  A 12-item scale that utilizes a 7-point Likert type scale with responses ranging from 1 (strongly disagree) to 7 (strongly agree). Total scores range from 12-84, with a higher score indicating higher mental health literacy.
Patient Activation: Patient Activation Measure (PAM) | 12 weeks
  13-item measure that assesses the patient's perception of their knowledge, skill, and confidence in self-management behavior. Scores range from 0-100, with a higher score indicating greater patient activation.
Effective Communication: Patients' Self-Competence Subscale (PSC) | 12 weeks
  A 16-item five point Likert scale that asks participants to rate items from 5 (important) to 1 (unimportant); a higher score indicates greater perceived self-competence and effective communication with a health care provider.
Symptom Severity: Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  A 14-item self-report measure that assesses anxiety and depression symptom severity. The HADS contains separate subscales (7 items each) for depression and anxiety; items are scored on a four point scale from 0-4, and a summative score is generated for each subscale. A cut score of 8 signifies an increased clinical risk for anxiety and depression.
Feasibility and Acceptability of Intervention | 12 weeks
  To assess feasibility, the frequency of refusals and incidence of complete intervention doses will be documented. Acceptability will be assessed by utilizing and adapted acceptability scale administered at the final time point.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa D Pinto-Foltz, PhD, RN, Principal Investigator — Case Western Reserve University
Locations (1):
- Frances Payne Bolton School of Nursing, Cleveland, Ohio, United States